CLINICAL TRIAL: NCT00219271
Title: Effect Of Zoledronic Acid On Circulating And Bone Marrow-Residing Prostate Cancer Cells In Patients With Clinically Localized Prostate Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: University of Athens (Other)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446GGR01
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; molecular staging; antitumor potential
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Zoledronic Acid

ARMS (1):
- Zoledronic acid (Experimental): 4 mg IV infused over 15 minutes every 3 months
  Interventions: Drug: Zoledronic acid

INTERVENTIONS:
Drug: Zoledronic acid

SUMMARY:
The objective of this study is to assess the effect Of zoledronic acid on circulating and bone marrow-residing prostate cancer cells in patients with clinically localized prostate cancer

ELIGIBILITY:
Inclusion Criteria

* Prostate cancer
* Radical prostatectomy or external beam irradiation therapy within 6 months before study entry.
* No bone metastases according to bone scan

Exclusion Criteria

* Metastatic prostate cancer
* Hormone ablation therapy for more than 3 months before/after radical prostatectomy and external beam irradiation therapy
* Treatment with bisphosphonates or other drugs known to affect the skeleton within the past year.

Other protocol-defined inclusion / exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2003-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To assess the activity of one year treatment with zoledronic acid | 12 mos

SECONDARY OUTCOMES:
Three-year disease free survival | 3 years
Change in bone mineral density at 12, 24 and 36 months versus baseline | 12, 24 and 36 months
Changes in bone resorption markers at 12, 24 and 36 months versus baseline | 12, 24 and 36 months
Safety and tolerability through abnormal values and AE reporting | upto 36 mos

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Athens, Greece

IPD SHARING:
Plan to Share IPD: No